CLINICAL TRIAL: NCT01215578
Title: A Multicenter Phase II Open Study Coupled With a Translational Assessment of Biomarkers Predictive of Response to Sunitinib in Patients With Poorly-differentiated Advanced/Inoperable NEURO-Endocrine Tumors.
Brief Title: Predictive Biomarkers of Response to Sunitinib in the Treatment of Poorly-differentiated NEURO-Endocrine Tumors
Acronym: NET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitement
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070145; 2007-005628-34 (EudraCT Number)
Record Dates: First submitted 2010-09-23; First posted 2010-10-06 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Neuroendocrine Tumors; Pancreatic Neoplasms; Advanced Disease; Sunitinib
Keywords: Neuroendocrine Tumors; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms, Nerve Tissue; Pancreatic Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Endocrine Gland Neoplasms; Adenoma, Islet Cell; Adenocarcinoma; Carcinoma; Adenoma; Digestive System Diseases; Pancreatic Diseases; Endocrine System Diseases; Sunitinib; Antineoplastic Agents; Therapeutic Uses; Pharmacologic Actions; Angiogenesis Inhibitors; Angiogenesis Modulating Agents; Growth Substances; Physiological Effects of Drugs; Growth Inhibitors
MeSH Terms: conditions — Neuroendocrine Tumors; Pancreatic Neoplasms; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms, Nerve Tissue; Digestive System Neoplasms; Neoplasms by Site; Endocrine Gland Neoplasms; Adenoma, Islet Cell; Adenocarcinoma; Carcinoma; Adenoma; Digestive System Diseases; Pancreatic Diseases; Endocrine System Diseases | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patient treated (Experimental): patient who receive sunitinib (SUTENT)
  Interventions: Drug: Sutent

INTERVENTIONS:
Drug: Sutent — sunitinib 37.5 mg/day (per os) for 6 months

SUMMARY:
The purpose of this study is to identify predictive molecular markers of response to continuous daily sunitinib at dose of 37.5 mg used in patients with poorly-differentiated Advanced/Inoperable NEURO-Endocrine Tumors.

Hypothesis:

* To distinguish molecular markers based on their expression at the initial biopsy, their detection by proteomic analysis and demonstrating that tumor or vascular cells are straightaway sensitive to sunitinib (markers sensitivity).
* The presence of these markers at the initial biopsy predict the sensitivity to sunitinib(Positive predictive value of markers)

DETAILED DESCRIPTION:
Neuroendocrine tumors (NET) are rare malignancies (1-2% of digestive cancers); and there is, in recent years, a slow but steady increase in their incidence. Despite the joint efforts of several research groups, which led to the new WHO classification (2002), the natural history of the disease remains heterogene and the resistance to conventional cytotoxic treatment remains the common denominator of these tumors.

Indeed, the prognosis of patients with metastatic disease remains poor despite numerous treatments (including: IFN, DTIC, 5-FU, doxorubicin, somatostatin analogues, etc.).

None of which showed a benefit in terms of survival. The main therapeutic objective is still to get a palliative effect on the symptoms and / or limit a few months tumor progression.

There are many publications showing that angiogenesis is one of the major mechanisms of tumor progression in TNE. But the multiple signaling pathways involved, the existence of alternative routes and their relationship to apoptosis inducing molecules remain unknown. Sunitinib is a new molecule in the family of tyrosine kinase inhibitors targeting multiple receptors which VEGFR, KIT, PDGF-R, FLT3 and RET. Since 2006 year, Sunitinib has been approved to treat advanced kidney cancer also called advanced renal cell carcinoma (a typically chemoresistant disease for which there was no active treatment available).

Many retrospective studies in patients showing that the TNE overexpress one or more targets of sunitinib. In Phase I trial, an antitumor activity has been identified in neuroendocrine tumors. In a phase II trial including 100 patients with well-differentiated TNE and carcinoids, sunitinib is associated with a response rate of 10%, and 82% of clinical benefit in the form of tumor stability.

Currently, an international randomised phase III trial initiated in well differentiated forms, but no studies are underway for poorly-differentiated TNE.

All of this suggests that sunitinib could represent an important therapeutic option for moderate, or poorly differentiated inoperable TNE and needs to be explored in this pathology by identifying predictive biomarkers of response.

ELIGIBILITY:
Inclusion Criteria:

* Digestive NET histopathologically proven, poorly-differentiated
* Inoperable/advanced NET (Tumor relapse inoperable or metastatic with no surgical indication).
* Tumor samples should be made available for analysis(diagnostic biopsy, surgical specimen)
* measurable disease defined by at least one lesion wich can be measured by at least one dimension :

  * equal or superior to 20 mm ( by conventional methods )
  * equal or superior to 10 mm (by spiral scan within 28 days before the beginning of the treatment)
* Performance status WHO ≤ 2.
* Adequate organ function :

  * hematology (absolute neutrophil count equal or superior to 1,5 x 10*9/l , platelet equal or superior to 100 x 10*9/l),
  * clearance of creatinine equal or superior to 60 ml/min),
  * AST/ALT ≤ 5 N, PAL ≤ 5 N, total bilirubin ≤ 2N.
* the selected women must be post-menopausal woman or surgically castrated or have to accept an effective contraception for the duration of the treatment and 3 month after.Women who are old enough to procreate must have a negative pregnancy test within the 72 hours of the beginning of the treatment.They must not be pregnant or to breastfeed.the selected men and theirs partners must be sterile or use an effective contraception for the duration of the treatment and 3 month after.

Exclusion Criteria:

* Hypersensitivity to sunitinib.
* Contraindication to sunitinib, including uncontrolled hypertension, medical history of cerebrovascular accident, unstable cardiac pathology despite optimal medical therapy (myocardial infarction within the 6 months prior to study drug administration, severe/unstable angina ), active hemorrhagic syndrome or concomitant treatment with anticoagulants.
* Any severe acute or chronic co-morbid that may compromise to comply with study participation: uncontrolled infection, symptomatic congestive heart failure, liver disturbance, chronic renal failure, active gastro-duodenal ulcer (nonexhaustive list).
* Known brain metastases.
* Diagnosis of any second malignancy within the last 3 years, except for basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri
* Current treatment on another clinical trial.
* Prior treatment with an investigational agent within 4 weeks.
* Prior treatment with intravenous biphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-10; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Predictive molecular markers of response to sunitinib | 1 year
  to assess the correlation between the expression of biomarkers and CT scan response. Patients are considered as responders when objective response (Partial or complete response) is showed on CT scan.

SECONDARY OUTCOMES:
The antitumor activity of sunitinib | 1 year
  * Objective response according to RECIST criteria (Time Frame: duration of study Safety issue: No).
  * Overall Survival (Time Frame: 6 months. Safety issue: No).
  * Progression-free survival (PFS)
  * Correlation between overall survival, PFS and tumor necrosis assessed on CT scan
Residual concentration | 2 months
  correlation between the concentration of sunitinib and its major active metabolite, SU012662, and objective response and /or toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Raymond, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, Hauts de Seine, France